CLINICAL TRIAL: NCT03347825
Title: A Retrospective Multi-Center Study for Evaluation of Clinical Outcomes With Lobectomy for Lung Cancer
Brief Title: Retrospective Multi-Center Study to Compare Perioperative Outcomes for Robotic-assisted Lobectomy With Those Associated With VATS and Open Lobectomy for Lung Cancer
Acronym: PORTaL
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVLob-001
Record Dates: First submitted 2017-10-31; First posted 2017-11-20 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Robotic-assisted lobectomy: Pre-operative, intra-operative and post-operative clinical, surgical and oncological information will be obtained from institutional records for patients who underwent robotic-assisted lobectomy for lung cancer.
  Interventions: Procedure: Robotic-assisted lobectomy using da Vinci Surgical System
- VATS (video assisted thoracic surgery) lobectomy: Pre-operative, intra-operative and post-operative clinical, surgical and oncological information will be obtained from institutional records for patients who underwent VATS lobectomy for lung cancer.
  Interventions: Procedure: VATS (video assisted thoracic surgery)
- Open lobectomy: Pre-operative, intra-operative and post-operative clinical, surgical and oncological information will be obtained from institutional records for patients who underwent open lobectomy for lung cancer.
  Interventions: Procedure: Open lobectomy

INTERVENTIONS:
Procedure: Robotic-assisted lobectomy using da Vinci Surgical System — Robotic-assisted lobectomy
  Groups: Robotic-assisted lobectomy
Procedure: VATS (video assisted thoracic surgery) — VATS (video assisted thoracic surgery)
  Groups: VATS (video assisted thoracic surgery) lobectomy
Procedure: Open lobectomy — Open lobectomy
  Groups: Open lobectomy

SUMMARY:
The main objective of this study is to evaluate and compare peri-operative outcomes of lobectomy compare with different approaches. The study aims to include patients with stage IA, IB, IIA, IIB and IIIA lung cancer that underwent lobectomy via robotic-assisted, VATS and open approach.

DETAILED DESCRIPTION:
This is a multi-center, retrospective chart review study of all consecutive lobectomies performed for clinical stage IA, IB, IIA, IIB and IIIA lung cancer, performed by participating surgeons at their respective institutions that meet all inclusion and exclusion criteria. All cases of lobectomy performed for clinical stages, IA, IB, IIA, IIB and IIIA lung cancer via robotic-assisted, VATS (video assisted thoracic surgery) and open approach that meet the study inclusion and exclusion criteria will be considered for inclusion in the study. The chart review and data collection will be performed in a reverse chronological order starting at 30 days prior to IRB approval of the study at the institution and going back to 2013 (i.e most current data in 2017 and chronologically going back through 2013). The retrospective chart review and data collection is anticipated to occur in two phases:

Baseline patient characteristics, perioperative and post-operative short term clinical and pathological outcomes data will be obtained from hospital records. Each participating institution will contribute approximately 100-800 cases from one or more surgeons. Since the data will have been de-identified, and is archival in nature, there will be no active subject recruitment and no patient consenting is required

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older
* Subject who has undergone elective robotic-assisted, VATS or open lobectomy for clinically diagnosed primary stage IA, IB, IIA, IIB and IIIA lung cancer, with or without neo-adjuvant therapy

Exclusion Criteria:

* Subject with stage IIIB lung cancer
* Subject who received lobectomy as an emergent procedure
* Subjects who received lobectomy for metastatic cancer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent robotic-assisted, VATS or open lobectomy for primary stage IA, IB, IIA, IIB and IIIA lung cancer, with or without neo-adjuvant therapy.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Chart review and data collection of clinical stage IB, IIA, IIB, IIIA cases | 2013-2019
  Compare peri-operative outcomes of robotic-assisted lobectomy with those associated with VATS and open lobectomy for lung cancer

CONTACTS AND LOCATIONS:
Locations (1):
- BaylorScott&White, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No